CLINICAL TRIAL: NCT05845814
Title: A Phase 1/2 Randomized, Umbrella Study to Evaluate the Safety and Efficacy of Pembrolizumab Plus Enfortumab Vedotin (EV) in Combination With Investigational Agents Versus Pembrolizumab Plus EV, as First-Line Treatment for Participants With Advanced Urothelial Carcinoma (KEYMAKER-U04): Substudy 04B
Brief Title: A Study of Efficacy and Safety of Pembrolizumab Plus Enfortumab Vedotin (EV) +/- Investigational Agents in First-Line Metastatic Urothelial Carcinoma (mUC) (MK-3475-04B/KEYMAKER-U04)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-04B; MK-3475-04B (Other: MSD); 2023-506385-30-00 (Registry Identifier: EU CT); U1111-1293-7564 (Registry Identifier: UTN); 2022-001371-14 (EudraCT Number)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Urothelial Carcinoma; Urothelial Neoplasms
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: In Part 1, participants will be randomized in a 1:1:1 ratio to receive either Arm A (coformulated favezelimab/pembrolizumab plus EV), Arm B (coformulated vibostolimab/pembrolizumab plus EV), or Arm C (pembrolizumab plus EV). If Part 2 is conducted, participants will be randomized in a 1:1:1 ratio to Arms A, B, and C or in a 1:1 ratio to Arms A and C or B and C, depending on the treatment arm(s) that are expanded in Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Coformulated favezelimab/pembrolizumab plus EV (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) as an intravenous (IV) infusion on Day 1 of every 3-week cycle for up to ~2 years (35 cycles) and EV at 1.25 mg/kg, administered as an IV infusion on Days 1 and 8 of every 3-week cycle until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Coformulated favezelimab/pembrolizumab; Combination Product: EV
- Arm B: Coformulated vibostolimab/pembrolizumab plus EV (Experimental): Participants will receive coformulated vibostolimab/pembrolizumab (200 mg/200 mg) as an IV infusion on Day 1 of every 3-week cycle, for up to ~2 years (35 cycles) and EV at 1.25 mg/kg, administered as an IV infusion on Days 1 and 8 of every 3-week cycle until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Coformulated vibostolimab/pembrolizumab; Combination Product: EV
- Arm C: Pembrolizumab plus EV (Active Comparator): Participants will receive 200 mg pembrolizumab as an IV infusion on Day 1 of every 3-week cycle for up to ~2 years (35 cycles) and EV at 1.25 mg/kg, administered as an IV infusion on Days 1 and 8 of every 3-week cycle, until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Combination Product: EV; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Coformulated favezelimab/pembrolizumab — Coformulated favezelimab/pembrolizumab (800 mg/200 mg) IV infusion
  Other Names: MK-4280A
  Arms: Arm A: Coformulated favezelimab/pembrolizumab plus EV
Biological: Coformulated vibostolimab/pembrolizumab — Coformulated vibostolimab/pembrolizumab (200 mg/200 mg) IV infusion
  Other Names: MK-7684A
  Arms: Arm B: Coformulated vibostolimab/pembrolizumab plus EV
Combination Product: EV — 1.25 mg/kg IV infusion
  Other Names: Padcev; ASG-22CE; ASG-22ME
Biological: Pembrolizumab — 200 mg IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm C: Pembrolizumab plus EV

SUMMARY:
This study is a substudy being conducted under one pembrolizumab umbrella master study KEYMAKER-U04. The substudy will consist of 2 parts. Part 1 will evaluate the efficacy and safety of coformulated favezelimab/pembrolizumab plus EV and coformulated vibostolimab/pembrolizumab plus EV relative to pembrolizumab plus EV. There will be no comparison of coformulated favezelimab/pembrolizumab plus EV versus coformulated vibostolimab/pembrolizumab plus EV. If ORR and/or DRR are substantially better on coformulated favezelimab/pembrolizumab plus EV and/or coformulated vibostolimab/pembrolizumab plus EV compared with pembrolizumab plus EV, after evaluation of the totality of data, the sponsor might consider Part 2 (expansion) to further characterize the efficacy and safety of the treatment arms under study.

DETAILED DESCRIPTION:
The master study for this substudy is MK-3475-U04/KEYMAKER-U04. The master study will not be screening any participants and will not be registered.

With Amendment 2, participants will discontinue treatment with coformulated vibostolimab/pembrolizumab (Arm B) and be transitioned to pembrolizumab only. Per protocol, no analysis of Part 2 primary or secondary outcome measures (including efficacy or safety) will occur since Part 2 of the study will no longer take place.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically documented, locally advanced/metastatic urothelial carcinoma (la/mUC).

  * Participants with mixed histology are eligible provided the urothelial component is ≥50% (and <10% plasmacytoid component)
  * Participants whose tumors contain any neuroendocrine component are not eligible (variant histology to be confirmed locally)
* Must not have received prior systemic therapy for la/mUC. The following therapies in earlier disease setting (eg, muscle-invasive urothelial carcinoma (MIUC)) are permitted:

  * Participants that received neoadjuvant or adjuvant chemotherapy are permitted.
  * Participants who received anti- programmed cell death 1 protein (PD-1) or programmed cell death ligand 1 (PD-L1) therapy for an earlier disease stage (eg, NMIBC, MIUC) with progression/recurrence >12 months from completion of therapy are permitted.
* Must provide an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion demonstrating UC, not previously irradiated, and adequate for biomarker evaluation. A newly obtained biopsy is strongly preferred, but not required if archival tissue is evaluable.
* Any AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Endocrine-related AEs adequately treated with hormone replacement or with <Grade 2 neuropathy are eligible.

Exclusion Criteria:

* Has a known additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy.
* Central nervous system (CNS) metastases are permitted on-study if all of the following are true: a) CNS metastases have been clinically stable for at least 4 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis; b) the participant is on a stable dose of ≤10 mg/day of prednisone or equivalent for at least 2 weeks (if requiring steroid treatment); c) participant does not have leptomeningeal disease.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention. Inhaled or topical steroids are permitted in the absence of active autoimmune disease. Physiologic replacement doses of corticosteroids are permitted for participants with adrenal insufficiency.
* Has active keratitis or corneal ulcerations. Superficial punctate keratitis is allowed if the disorder is being adequately treated in the opinion of the investigator.
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy.
* Has a history of uncontrolled diabetes.
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection (viral, bacterial, or fungal) requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has hepatitis B or hepatitis C virus infection.
* Has had major surgery within 4 weeks prior to first dose of study intervention.
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Objective Response Rate (ORR) | Up to ~4 years
  ORR is defined as the percentage of participants who achieve a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR). ORR will be reported for participants in Part 1.
Part 1: Percentage of Participants experiencing an Adverse Event (AE) | Up to ~4 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants experiencing an AE in Part 1 will be reported.
Part 1: Percentage of Participants who Discontinue study interventions due to an AE | Up to ~4 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinue study interventions due to an AE in Part 1 will be reported.
Part 1: Percentage of Participants with Dose-limiting toxicities (DLT) | Up to 21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0). The number of participants who experience a DLT in Part 1 will be reported.
Part 2: Progression Free Survival (PFS) | Up to ~4 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. PFS will be reported for participants in Part 2.

SECONDARY OUTCOMES:
Part 1: PFS | Up to ~4 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. PFS will be reported for participants in Part 1.
Part 1: Duration of Response (DOR) | Up to ~4 years
  For participants who demonstrate confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR will be reported for participants in Part 1.
Part 2: Overall Survival (OS) | Up to ~4 years
  OS is defined as the time from randomization to death due to any cause. OS will be reported for participants in Part 2.
Part 2: ORR | Up to ~4 years
  ORR is defined as the percentage of participants who achieve a confirmed CR or PR per RECIST 1.1 as assessed by BICR. ORR will be reported for participants in Part 2.
Part 2: DOR | Up to ~4 years
  For participants who demonstrate confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR will be reported for participants in Part 2.
Part 2: Percentage of Participants experiencing an Adverse Event (AE) | Up to ~4 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants experiencing an AE in Part 2 will be reported.
Part 2: Percentage of Participants who Discontinue study interventions due to an AE | Up to ~4 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinue study interventions due to an AE in Part 2 will be reported.
Part 2: Percentage of Participants with Dose-limiting toxicities (DLT) | Up to 21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0). The number of participants who experience a DLT in Part 2 will be reported.
Part 1: Mean Change from baseline in the global health status/quality of life of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLC-C30) (Items 29 and 30) | Baseline and up to ~4 years
  Participants are asked to answer questions 29 and 30 from the EORTC QLC-C30. Questions 29 and 30 use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 1.
Part 1: Mean Change from baseline in the physical functioning scale of the EORTC QLQ-C30 | Baseline and up to ~4 years
  Participants are asked to answer questions about their physical functioning from the EORTC QLC-C30. These questions use a 4-point scale (1=not at all to 4=very much) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 1.
Part 1: Mean Change from Baseline in the European Quality of Life 5 Dimensions, 5-level Questionnaire (EQ-5D-5L) visual analog score (VAS) | Baseline and up to ~4 years
  The EQ-5D-5L is a descriptive five-dimensional system of evaluation. The five dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants rate each dimension on 5 levels ranging from 1 (no problems) to 5 (extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale on which the participant rates their general state of health. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 1.
Part 2: Mean Change from baseline in the global health status/quality of life of the EORTC QLC-C30 (Items 29 and 30) | Baseline and up to ~4 years
  Participants are asked to answer questions 29 and 30 from the EORTC QLC-C30. Questions 29 and 30 use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 2.
Part 2: Mean Change from baseline in the physical functioning scale of the EORTC QLQ-C30 | Baseline and up to ~4 years
  Participants are asked to answer questions about their physical functioning from the EORTC QLC-C30. These questions use a 4-point scale (1=not at all to 4=very much) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 2.
Part 2: Mean Change from Baseline in the EQ-5D-5L visual analog score (VAS) | Baseline and up to ~4 years
  The EQ-5D-5L is a descriptive five-dimensional system of evaluation. The five dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants rate each dimension on 5 levels ranging from 1 (no problems) to 5 (extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale on which the participant rates their general state of health. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. The mean change from baseline will be reported for Part 2.
Part 1: Time-to-Deterioration (TTD) for the global health status/quality of life of the EORTC QLQ-C30 (Items 29 and 30) | Up to ~4 years
  Participants are asked to answer questions 29 and 30 from the EORTC QLC-C30. Questions 29 and 30 use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. TTD is defined as the time from the first GHS/QoL assessment to deterioration (defined as ≥10-point decrease in GHS/QoL score from baseline) or death, whichever occurs first. The TTD in GHS/QoL score of participants will be reported for Part 1.
Part 1: TTD for the physical functioning scale of the EORTC QLQ-C30 | Up to ~4 years
  Participants are asked to answer questions about their physical functioning from the EORTC QLC-C30. These questions use a 4-point scale (1=not at all to 4=very much) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. TTD is defined as the time from the first GHS/QoL assessment to deterioration (defined as ≥10-point decrease in GHS/QoL score from baseline) or death, whichever occurs first. The TTD in GHS/QoL score of participants will be reported for Part 1.
Part 1: TTD for the EQ-5D-5L VAS | Up to ~4 years
  The EQ-5D-5L is a descriptive five-dimensional system of evaluation. The five dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants rate each dimension on 5 levels ranging from 1 (no problems) to 5 (extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale on which the participant rates their general state of health. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. TTD is defined as the time from the first EQ-5D-5L VAS assessment to deterioration (defined as ≥7-point decrease in EQ-5D-5L VAS score more from baseline) or death, whichever occurs first. The TTD in EQ-5D-5L VAS score of participants will be reported for Part 1.
Part 2: TTD for the global health status/quality of life of the EORTC QLQ-C30 (Items 29 and 30) | Up to ~4 years
  Participants are asked to answer questions 29 and 30 from the EORTC QLC-C30. Questions 29 and 30 use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. TTD is defined as the time from the first GHS/QoL assessment to deterioration (defined as ≥10-point decrease in GHS/QoL score from baseline) or death, whichever occurs first. The TTD in GHS/QoL score of participants will be reported for Part 2.
Part 2: TTD for the physical functioning scale of the EORTC QLQ-C30 | Up to ~4 years
  Participants are asked to answer questions about their physical functioning from the EORTC QLC-C30. These questions use a 4-point scale (1=not at all to 4=very much) to evaluate overall health and quality of life. Scores were transformed to a range of 0 to 100 using a standard EORTC algorithm. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. TTD is defined as the time from the first GHS/QoL assessment to deterioration (defined as ≥10-point decrease in GHS/QoL score from baseline) or death, whichever occurs first. The TTD in GHS/QoL score of participants will be reported for Part 2.
Part 2: TTD for the EQ-5D-5L VAS | Up to ~4 years
  The EQ-5D-5L is a descriptive five-dimensional system of evaluation. The five dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants rate each dimension on 5 levels ranging from 1 (no problems) to 5 (extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale on which the participant rates their general state of health. Negative change from baseline values indicated deterioration in health status or functioning and positive changes indicated improvement. TTD is defined as the time from the first EQ-5D-5L VAS assessment to deterioration (defined as ≥7-point decrease in EQ-5D-5L VAS score more from baseline) or death, whichever occurs first. The TTD in EQ-5D-5L VAS score of participants will be reported for Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (47):
- United States (14):
  - Moores Cancer Center ( Site 3028), La Jolla, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 3045), Orange, California
  - UCSF Medical Center at Mission Bay ( Site 3044), San Francisco, California
  - Anschutz Cancer Pavilion ( Site 3017), Aurora, Colorado
  - Emory University School of Medicine ( Site 3043), Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 3011), Indianapolis, Indiana
  - Dana-Farber Cancer Institute ( Site 3047), Boston, Massachusetts
  - Siteman Cancer Center ( Site 3038), St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai ( Site 3018), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 3031), New York, New York
  - Duke Cancer Institute ( Site 3027), Durham, North Carolina
  - Cleveland Clinic-Taussig Cancer Center ( Site 3036), Cleveland, Ohio
  - UPMC Hillman Cancer Center ( Site 3014), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute-HCI Clinical Trials Office ( Site 3041), Salt Lake City, Utah
- Australia (2):
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 3951), Brisbane, Queensland
  - Austin Health-Cancer Clinical Trials Centre ( Site 3950), Heidelberg, Victoria
- Canada (3):
  - The Ottawa Hospital - General Campus-The Ottawa Hospital Cancer Centre ( Site 3105), Ottawa, Ontario
  - Sunnybrook Research Institute - Odette Cancer Centre ( Site 3108), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 3106), Toronto, Ontario
- Chile (4):
  - FALP-UIDO ( Site 3151), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 3155), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 3158), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 3152), Antofagasta
- France (5):
  - CHU de Bordeaux Hop St ANDRE ( Site 3607), Bordeaux, Aquitaine
  - Centre Georges François Leclerc-Centre de recherche clinique ( Site 3608), Dijon, Cote-d Or
  - Oncopole Claudius Regaud ( Site 3610), Toulouse, Haute-Garonne
  - centre hospitalier lyon sud ( Site 3606), Pierre-Bénite, Rhone
  - Hôpital Européen Georges Pompidou ( Site 3605), Paris
- Israel (3):
  - Rambam Health Care Campus-Oncology Division ( Site 3501), Haifa
  - Rabin Medical Center-Oncology ( Site 3504), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 3503), Ramat Gan
- Italy (3):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 3406), Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 3405), Milan, Lombardy
  - Ospedale San Raffaele-Oncologia Medica ( Site 3403), Milan
- Netherlands (3):
  - Maastricht UMC+ ( Site 3304), Maastricht, Limburg
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL)-medical oncology ( Site 3302), Amsterdam, North Holland
  - Erasmus Medisch Centrum-Medical Oncology ( Site 3303), Rotterdam, South Holland
- South Korea (3):
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 3903), Seoul
  - Asan Medical Center-Department of Oncology ( Site 3901), Seoul
  - Samsung Medical Center ( Site 3902), Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron ( Site 3767), Barcelona, Catalonia
  - Hospital Clinico San Carlos ( Site 3765), Madrid
- Taiwan (3):
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 3802), Kaohsiung City
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 3803), Tainan
  - National Taiwan University Hospital-Oncology ( Site 3801), Taipei
- United Kingdom (2):
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 3206), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 3201), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26285&tenant=MT_MSD_9011